CLINICAL TRIAL: NCT03769129
Title: A Prospective，Single Center, Randomized Control，Phase III Clinical Study for Evaluating the Safety and Efficacy of Pembrolizumab Combined With MWA for Patients With Stage ⅢB-Ⅳ NSCLC Who Failed With First-line Therapy
Brief Title: Evaluating the Safety and Efficacy of Pembrolizumab Combined With MWA for Advanced NSCLC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZZWMAICI-005
Record Dates: First submitted 2018-11-12; First posted 2018-12-07 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Microwave ablation; Pembrolizumab; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microwave ablation (Experimental): Firstly, microwave ablation performed at our department by interventional radiologist, then Pembrolizumab will be administered at a dose of 2 mg/kg every three weeks.
  Interventions: Drug: Pembrolizumab; Procedure: microwave ablation
- Pembrolizumab (Other): Firstly, pembrolizumab was administered intravenously at a dose of 2 mg/kg. Then microwave ablation will be performed if there is no immune-related adverse reactions. Pembrolizumab will also be continuously administered every three weeks until the imaging evaluation of the disease progress.
  Interventions: Drug: Pembrolizumab; Procedure: microwave ablation

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab
  Other Names: Keytruda
Procedure: microwave ablation — microwave ablation

SUMMARY:
This is a prospective, randomized, single clinical study designed to evaluate its safety and efficacy by using Microwave Ablation combine with Pembrolizumab in patients with Stage ⅢB-Ⅳ Non-small Cell Lung.Cancer (NSCLC) who failed with first-line therapy.

DETAILED DESCRIPTION:
Lung cancer is one of the most common malignant tumors in the world and has become the No. 1 cause of death from malignant tumors in China. Non-small cell lung cancer (NSCLC) includes squamous cell carcinomas, adenocarcinomas, and large cell carcinomas and accounts for about 80-85% of all lung cancers. NSCLC cancer cells divide slowly in a diffusive manner and metastasize at a relatively late stage compared to small cell carcinomas. A majority of patients with NSCLC are already in advanced stages and have a low 5-year survival rate.

Treatments for advanced NSCLC include chemotherapy ,targeted therapies and immunotherapy. The microwave ablation is the good choice for patients who cannot tolerate surgical resection. A large number of studies have shown that local minimally invasive ablation therapy within a certain temperature range can stimulate the body to produce an immune response to varying degrees. The study found that for a variety of malignant tumor models, thermal ablation local treatment of in situ tumors, while the disappearance of other metastatic lesions, and treated mice are resistant to secondary vaccination of the same tumor, proving that thermal ablation therapy stimulates long-lasting Anti-tumor immunity. Pembrolizumab are representative drugs for immunosuppressive agents, and its indications have been approved in various types of tumors, including advanced melanoma, advanced squamous non-small cell lung cancer, advanced renal cell carcinoma, and classical Hodgkin's lymphoma and late recurrent head and neck squamous cell carcinoma patients. Whether the combination of the two can cause a stronger anti-tumor immune response in the body. However, the flexibility, safety and efficacy of using Microwave Ablation combine with Pembrolizumab in NSCLC patients are still unclear.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed IIIB or IV non-small cell lung cancer.
2. Previously accepted first-line standard treatment failure or recurrence
3. At least one measurable lesion.
4. The patient has not received any other anti-cancer treatment within four weeks.
5. Any gender, age ≥18 years
6. ECOG PS : 0-2 points
7. Expected survival ≥ 6 months
8. The level of organ function meets the following criteria.

(1) subject to the standard blood test: ANC ≥ 1.5×109 / L, PLT ≥ 50×109 / L, Hb ≥ 90g/L.

(2) biochemical tests must meet the following criteria: TBIL<1.5×ULN, ALT, AST <2.5×ULN ( if liver metastasis ALT, AST can be <5×ULN), BUN, and Cr ≤ 1×ULN).

9. Female patients in child bearing period must have evidence of negative pregnancy test, and agree to take effective contraceptive measures until 6months after therapy.

10. Subjects volunteered to join the study, signed informed consent, good compliance, with follow-up.

Exclusion Criteria:

1. Patients with two or more kinds of tumors.
2. Patients with active viral or bacterial infection, and have failed to be controlled by anti-infective treatment.
3. Patients with seropositive response of Human immunodeficiency virus (HIV) and syphilis, or fail to control the hepatitis B virus or hepatitis C virus infection.
4. Patients with active rheumatic diseases, organ transplantation and other diseases affecting the immune system seriously.
5. Patients with severe heart and lung dysfunction.
6. Patients with severe chronic diseases of kidney, liver and other important organs.
7. Patients with any other serious illness that the investigators consider it will may affect the patient's treatments, follow-up or assessment, including any uncontrolled clinically significant neurological or psychiatric disorders, immunoregulatory diseases, metabolic diseases, infectious diseases and so on.
8. Patients who take part in clinical trials of other drugs or biological therapy at present or within 30 days before enrollment.
9. Patients who need long-term use of immunosuppressive drugs or patients who are undergoing treatment of autoimmune diseases.
10. Patients who need long-term use of glucocorticoid.
11. Women patients in gestation period or suckling period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  Overall survival (OS) will be defined as the elapsed time from the enrollment to death from any cause. For surviving patients, follow-up will be censored at the date of last contact (or last date known to be alive). Follow-up for OS will occur every 12 weeks (±1 month) until death or withdrawal of consent from the study.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events（Safety） | 2 years
  All the local reactions, systemic reactions, all the adverse events and serious adverse events obtained during the study of all the patients included in the first stage and the second stage of this study
Progression-Free Survival | 2 years
  From enrollment to progression of disease.

CONTACTS AND LOCATIONS:
Overall Officials: zhang zhenfeng, MD,PHD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- zhang Zhenfeng, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Don not plan